CLINICAL TRIAL: NCT01027871
Title: A Phase 2 Study of LY2605541 Compared With Insulin Glargine in the Treatment of Type 2 Diabetes Mellitus
Brief Title: A Study for Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12149; I2R-MC-BIAC (Other: Eli Lilly and Company)
Record Dates: First submitted 2009-12-08; First posted 2009-12-09 (Estimated); Results first posted 2018-06-08 (Actual); Last update posted 2018-06-08 (Actual); Status verified 2018-05

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — LY2605541; Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- LY2605541 Dosing Algorithm 1 (Experimental): Participants took both LY2605541 and their pre-study insulin for first several days
  Interventions: Drug: LY2605541
- LY2605541 Dosing Algorithm 2 (Experimental): Participants took only LY2605541 with first dose doubled
  Interventions: Drug: LY2605541
- Insulin glargine (Active Comparator)
  Interventions: Drug: insulin glargine

INTERVENTIONS:
Drug: LY2605541 — subcutaneous injection of LY2605541 every morning with dose titration based on blood glucose measures for 12 weeks
  Arms: LY2605541 Dosing Algorithm 1; LY2605541 Dosing Algorithm 2
Drug: insulin glargine — subcutaneous injection of insulin glargine every morning with dose titration based on blood glucose measures for 12 weeks
  Arms: Insulin glargine

SUMMARY:
Comparison of fasting blood glucose levels in patients with Type 2 diabetes after 12 weeks of treatment with a new basal insulin analog or with insulin glargine.

DETAILED DESCRIPTION:
Patients in this study will continue to use their stable prestudy dose of metformin and/or a sulfonylurea. Prestudy therapy also includes once daily insulin glargine or neutral protamine Hagedorn (NPH) insulin. The 12-week active treatment phase will be followed by a 4-week follow-up period, during which patients will return to the basal insulin recommended by the investigator.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus (T2DM) for at least 1 year
* At least 18 years of age
* Using metformin and/or sulfonylurea(s) with once daily glargine or NPH for at least 3 months prior to the study. Prestudy dose requirements: insulin dose maximum 1.0 unit/kilogram/day (U/kg/day). Oral antihyperglycemic medications (OAMs): Metformin dose at least 1500 milligram/day (mg/day) and/or sulfonylurea dose at least half the maximum daily dose specified in the local package insert. OAM doses stable for 6 weeks prior to the study.
* Hemoglobin A1c (HbA1c) less than or equal to 10.5% before randomization
* Body Mass Index (BMI) 19 to 45 kilogram/square meter (kg/m²)
* Capable and willing to prepare and inject insulin with a syringe while continuing to use the prestudy OAMs, monitor own blood glucose; complete the study diary; be receptive to diabetes education; comply with study visits and receive telephone calls between visits
* Women of childbearing potential must test negative for pregnancy before receiving treatment and agree to use reliable birth control until completing the follow-up visit

Exclusion Criteria:

* Long-term use of short- or rapid-acting or premixed insulin within the 6 months before the study. Short-term insulin therapy or occasional use are permitted
* Use of any glucose-lowering medications not allowed by the inclusion criteria in the 3 months before entry into the study
* Use of prescription or over-the-counter medications to promote weight loss within 3 months before entry into the study
* Current participation in a weight loss program, or plans to do so during the study
* Treatment with any antibody-based therapy within 6 months prior to the study
* Use of chronic (>14 consecutive days) systemic glucocorticoid therapy currently or within 4 weeks prior to the study
* More than 1 episode of severe hypoglycemia within 6 months prior to the study, or currently diagnosed with hypoglycemia unawareness
* 2 or more emergency room visits or hospitalizations due to poor glucose control in the 6 months preceding the study
* Liver disease
* History of renal transplantation, current renal dialysis, or creatinine >2.0 milligram/deciliter (mg/dL) (177 micromole/Liter [μmol]/L)
* Cardiac disease with a marked impact on physical functioning
* Clinically significant electrocardiogram (ECG) abnormalities at screening
* Malignancy other than basal cell or squamous cell skin cancer
* Fasting triglycerides >500 mg/dL
* Known diabetic autonomic neuropathy
* Known hypersensitivity or allergy to study insulin or its excipients
* Blood transfusion or severe blood loss within 3 months prior to entry into the study or known hemoglobinopathy, hemolytic anemia, or sickle cell anemia, or any other traits of hemoglobin abnormalities known to interfere with the HbA1c methodology
* Irregular sleep/wake cycle
* Women who are breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 289 (Actual)
Dates: Start 2010-01; Primary Completion 2010-12 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (25):
- United States (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Idaho Falls, Idaho
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Minneapolis, Minnesota
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dallas, Texas
- Australia (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Coffs Harbour, New South Wales
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Keswick, South Australia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ringwood East, Victoria
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fremantle, Western Australia
- Hungary (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Budapest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gyula
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Veszprém
- Poland (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bialystok
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lublin
- Puerto Rico (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hato Rey, San Juan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Manatí
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Juan
- Romania (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cluj-Napoca
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Iași
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Târgu Mureş
- Russia (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Arkhangelsk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Moscow
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rostov-on-Don
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint Petersburg
- Spain (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Alicante
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dos Hermanas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Málaga

REFERENCES:
- [Background] Workgroup on Hypoglycemia, American Diabetes Association. Defining and reporting hypoglycemia in diabetes: a report from the American Diabetes Association Workgroup on Hypoglycemia. Diabetes Care. 2005 May;28(5):1245-9. doi: 10.2337/diacare.28.5.1245. No abstract available. PMID 15855602
- [Derived] Qu Y, White RD, Ruberg SJ. Accurate Collection of Reasons for Treatment Discontinuation to Better Define Estimands in Clinical Trials. Ther Innov Regul Sci. 2023 May;57(3):521-528. doi: 10.1007/s43441-022-00491-0. Epub 2022 Dec 21. PMID 36542287
- [Derived] Bergenstal RM, Rosenstock J, Bastyr EJ 3rd, Prince MJ, Qu Y, Jacober SJ. Lower glucose variability and hypoglycemia measured by continuous glucose monitoring with novel long-acting insulin LY2605541 versus insulin glargine. Diabetes Care. 2014;37(3):659-65. doi: 10.2337/dc12-2621. Epub 2013 Nov 6. PMID 24198302
- [Derived] Bergenstal RM, Rosenstock J, Arakaki RF, Prince MJ, Qu Y, Sinha VP, Howey DC, Jacober SJ. A randomized, controlled study of once-daily LY2605541, a novel long-acting basal insulin, versus insulin glargine in basal insulin-treated patients with type 2 diabetes. Diabetes Care. 2012 Nov;35(11):2140-7. doi: 10.2337/dc12-0060. Epub 2012 Oct 9. PMID 22787177

RESULTS

PARTICIPANT FLOW:
Groups:
- LY2605541 Algorithm 1: Participants took both LY2605541 and their pre-study insulin for first several days
- LY2605541 Algorithm 2: Participants took only LY2605541 with first dose doubled
Period: Overall Study
Arm/Group | Insulin Glargine | LY2605541 Algorithm 1 | LY2605541 Algorithm 2
Started | 93 | 98 | 98
Received at Least One Dose of Study Drug | 93 | 98 | 97
Completed | 91 | 85 | 91
Not Completed | 2 | 13 | 7
Not completed — Physician Decision | 1 | 5 | 0
Not completed — Protocol Violation | 0 | 2 | 2
Not completed — Withdrawal by Subject | 1 | 2 | 2
Not completed — Adverse Event | 0 | 2 | 2
Not completed — Sponsor Decision | 0 | 2 | 0
Not completed — Discontinued Prior to Treatment | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least one dose of study drug.
Groups:
- LY2605541 Algrithm 2: Participants took only LY2605541 with first dose doubled
- Total: Total of all reporting groups
Arm/Group | Insulin Glargine | LY2605541 Algorithm 1 | LY2605541 Algrithm 2 | Total
Number analyzed (Participants) | 93 | 98 | 97 | 288
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.74 (7.94) | 58.57 (9.99) | 59.23 (9.28) | 59.49 (9.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 41 | 48 | 135
  Male | 47 | 57 | 49 | 153
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 0 | 4 | 2 | 6
  Black or African American | 4 | 2 | 6 | 12
  Multiple | 1 | 0 | 0 | 1
  White | 87 | 0 | 0 | 87
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 23 | 31 | 37 | 91
  Hungary | 5 | 5 | 6 | 16
  Puerto Rico | 12 | 8 | 9 | 29
  Poland | 0 | 2 | 2 | 4
  Spain | 13 | 11 | 12 | 36
  Romania | 12 | 13 | 12 | 37
  Australia | 10 | 5 | 6 | 21
  Russia | 18 | 13 | 12 | 43

OUTCOME MEASURES:

1. Primary Outcome: Fasting Blood Glucose (FBG) Level at Week 12 Endpoint as Measured by the 8-Point Self-Monitored Blood Glucose (SMBG) Profiles
Description: 8-point SMBG profiles are measured at morning FBG, midday and evening pre-meal blood glucose (BG), 2-hour postprandial BG after each of the 3 main meals, bedtime BG, 0300 hours BG. Least squares (LS) mean of the FBG is from mixed-model repeated measures (MMRM) approach, which includes fixed effects of treatment (LY2605541 algorithm 1 and 2, glargine); dose conversion (pre-interim analysis [IA], post-IA); stratification variables (country, baseline daily basal insulin dose group, and baseline hemoglobin A1c [HbA1c] group); visit; visit and treatment interaction; random effect for participant.
Time Frame: Week 12
Population: All randomized participants who took at least one dose of study drug with non-missing baseline value and at least one non-missing post-baseline value.
Measure: Least Squares Mean (Standard Error); unit: millimoles per Liter (mmol/L)
Groups:
- LY2605541 Algorithm 1: Participants took both LY2605541 and their pre-study insulin for first several days
  Subcutaneous injection of LY2605541 every morning with dose titration based on blood glucose measures for 12 weeks
- LY2605541 Algorithm 2: Participants took only LY2605541 with first dose doubled
  Subcutaneous injection of LY2605541 every morning with dose titration based on blood glucose measures for 12 weeks
Arm/Group | Insulin Glargine | LY2605541 Algorithm 1 | LY2605541 Algorithm 2
Number analyzed (Participants) | 89 | 86 | 91
millimoles per Liter (mmol/L) | 6.83 (0.22) | 7.15 (0.22) | 6.84 (0.22)
Statistical Analysis 1: Comparison: Insulin Glargine vs LY2605541 Algorithm 2; Test type: Superiority or Other; p = 0.433, Mixed Models Analysis — The statistical significance level is 0.10; Least Squares Mean Difference (Final) = 0.17, 90% CI 2-sided [-0.18 to 0.52] — The Least Squares Mean Difference = LY Combined - Insulin Glargine; and 90% confidence interval (CI) = 90% CI of the least squares mean difference

2. Secondary Outcome: Change From Baseline in Fasting Blood Glucose (FBG) at Week 12 Endpoint
Description: FBG is measured by 8-point SMBG profiles, which are measured at morning FBG, midday pre-meal BG, evening pre-meal BG, 2-hour postprandial BG after each of the 3 main meals, bedtime BG, 0300 hours BG. LS mean of the change from baseline to 12 weeks is from MMRM approach, which includes fixed effects of treatment (LY2605541 algorithm 1 and 2, glargine); dose conversion (pre-IA, post-IA); stratification variables (country, baseline daily basal insulin dose group, and baseline HbA1c group); visit; visit and treatment interaction; and random effect for participant.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmol/Liter
Groups:
- LY2605541 Combined: LY2605541 Dosing Algorithm 1 + LY2605541 Dosing Algorithm 2
  Algorithm 1: Participants took both LY2605541 and their pre-study insulin for first several days
  Algorithm 2: Participants took only LY2605541 with first dose doubled
  Subcutaneous injection of LY2605541 every morning with dose titration based on blood glucose measures for 12 weeks
Arm/Group | Insulin Glargine | LY2605541 Combined
Number analyzed (Participants) | 89 | 177
mmol/Liter | -1.77 (0.26) | -1.97 (0.21)
Statistical Analysis 1: Comparison: Insulin Glargine; Test type: Superiority or Other; p = 0.388, Mixed Models Analysis — The statistical significance level is 0.10; Least Squares Mean Difference (Final) = -0.20, 90% CI 2-sided [-0.59 to 0.19] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Change From Baseline in Hemoglobin A1c (HbA1c) at Week 12 Endpoint
Description: HbA1c is a form of hemoglobin which is measured primarily to identify the average plasma glucose concentration over prolonged periods of time. LS mean of the change from baseline is from MMRM approach. MMRM model includes fixed effects of treatment (LY2605541 dose algorithm 1 and 2, glargine); dose conversion (pre-IA, post-IA); stratification variables (country, baseline daily basal insulin dose group); baseline HbA1c; visit; visit and treatment interaction; and a random effect for participant.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage of glycated hemoglobin
Arm/Group | Insulin Glargine | LY2605541 Combined
Number analyzed (Participants) | 91 | 176
percentage of glycated hemoglobin | -0.64 (0.08) | -0.74 (0.06)
Statistical Analysis 1: Comparison: Insulin Glargine vs LY2605541 Combined; Test type: Superiority or Other; p = 0.197, Mixed Models Analysis — The statistical significance level is 0.10; Least Squares Mean Difference (Final) = -0.09, 90% CI 2-sided [-0.21 to 0.03] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Percentage of Participants With HbA1c <7.0% and ≤6.5% at Week 12 Endpoint
Description: HbA1c is a form of hemoglobin which is measured primarily to identify the average plasma glucose concentration over prolonged periods of time.
Time Frame: Week 12
Population: All randomized participants who took at least one dose of study drug, last observation carried forward (LOCF). Arms are combined due to
Measure: Number; unit: percentage of participants
Groups:
- LY2605541 Combined: Algorithm 1: Participants took both LY2605541 and their pre-study insulin for first several days Algorithm 2: Participants took only LY2605541 with first dose doubled Subcutaneous injection of LY2605541 every morning with dose titration based on blood glucose measures for 12 weeks
Arm/Group | Insulin Glargine | LY2605541 Combined
Number analyzed (Participants) | 91 | 183
percentage of participants
  HbA1c <7.0% | 48.4 | 51.9
  HbA1c ≤6.5% | 23.1 | 29.5
Statistical Analysis 1: Comparison: Insulin Glargine vs LY2605541 Combined; Test type: Superiority or Other; p = 0.609, Fisher Exact — The statistical significance level is 0.10. P-value is for HbA1c <7.0%
Statistical Analysis 2: Comparison: Insulin Glargine vs LY2605541 Combined; Test type: Superiority or Other; p = 0.314, Fisher Exact — The statistical significance level is 0.10. P-value is for HbA1c ≤6.5%

5. Secondary Outcome: Percentage of Participants With HbA1c <7.0% and HbA1c ≤6.5% at Week 12 Endpoint Who Did Not Experience a Hypoglycemic Episode During Treatment
Description: HbA1c is a form of hemoglobin which is measured primarily to identify the average plasma glucose concentration over prolonged periods of time. Hypoglycemia episode is defined as any time a participant feels that he/she is experiencing a sign or symptom that is associated with hypoglycemia or has a BG level of ≤3.9 millimole/Liter (mmol/L) (≤70 milligram/deciliter [mg/dL]) even if it was not associated with signs, symptoms, or treatment (consistent with current guidelines [ADA 2005]).
Time Frame: Week 12
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Insulin Glargine | LY2605541 Combined
Number analyzed (Participants) | 92 | 188
percentage of participants
  HbA1c <7.0% | 11.96 | 16.49
  HbA1c ≤6.5% | 6.52 | 7.98
Statistical Analysis 1: Comparison: Insulin Glargine vs LY2605541 Combined; Test type: Superiority or Other; p = 0.375, Fisher Exact — The statistical significance level is 0.10. P-value is for HbA1c <7.0%
Statistical Analysis 2: Comparison: Insulin Glargine vs LY2605541 Combined; Test type: Superiority or Other; p = 0.811, Fisher Exact — The statistical significance level is 0.10. P- value is for HbA1c ≤6.5%

6. Secondary Outcome: 8-Point Self-Monitored Blood Glucose (SMBG) Measures at Week 12 Endpoint
Description: 8-point SMBG profiles are measured at morning FBG, midday pre-meal BG, evening pre-meal BG, 2-hour postprandial BG after each of the 3 main meals, bedtime BG, 0300 hours BG. LS mean is obtained using MMRM approach, which includes fixed effects of treatment (LY2605541 algorithm 1 and 2, glargine); dose conversion (pre-IA, post-IA); stratification variables (country, baseline daily basal insulin dose group, and baseline HbA1c group); visit; visit and treatment interaction; and a random effect for participant.
Time Frame: Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Insulin Glargine | LY2605541 Combined
Number analyzed (Participants) | 92 | 191
mmol/L
  Morning 2-hr postprandial BG: number analyzed (Participants) | 87 | 175
  Morning 2-hr postprandial BG | 9.54 (0.31) | 9.11 (0.25)
  Midday Pre-meal BG: number analyzed (Participants) | 89 | 176
  Midday Pre-meal BG | 7.47 (0.28) | 7.23 (0.23)
  Midday 2-hr postprandial BG: number analyzed (Participants) | 88 | 175
  Midday 2-hr postprandial BG | 9.49 (0.28) | 9.22 (0.22)
  Evening Pre-meal BG: number analyzed (Participants) | 89 | 176
  Evening Pre-meal BG | 7.92 (0.28) | 7.80 (0.22)
  Evening 2-hr postprandial BG: number analyzed (Participants) | 89 | 176
  Evening 2-hr postprandial BG | 9.99 (0.30) | 9.74 (0.24)
  Bed time BG: number analyzed (Participants) | 80 | 160
  Bed time BG | 9.44 (0.31) | 9.15 (0.25)
  0300 hours BG: number analyzed (Participants) | 89 | 170
  0300 hours BG | 7.26 (0.25) | 7.36 (0.20)
Statistical Analysis 1: Comparison: Insulin Glargine vs LY2605541 Combined; Test type: Superiority or Other; p = 0.144, Mixed Models Analysis — The statistical significance level is 0.10. P- value is for morning 2-hr postprandial BG; Least Squares Mean Difference (Final) = -0.43, 90% CI 2-sided [-0.92 to 0.05] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Insulin Glargine vs LY2605541 Combined; Test type: Superiority or Other; p = 0.360, Mixed Models Analysis — The statistical significance level is 0.10. P-value is for midday pre-meal BG; Least Squares Mean Difference (Final) = -0.25, 90% CI 2-sided [-0.70 to 0.20] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Insulin Glargine vs LY2605541 Combined; Test type: Superiority or Other; p = 0.342, Mixed Models Analysis — The statistical significance level is 0.10. P-value is for midday 2-hr postprandial BG; Least Squares Mean Difference (Final) = -0.26, 90% CI 2-sided [-0.72 to 0.19] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Insulin Glargine vs LY2605541 Combined; Test type: Superiority or Other; p = 0.654, Mixed Models Analysis — The statistical significance level is 0.10. P-value is for evening pre-meal BG; Least Squares Mean Difference (Final) = -0.12, 90% CI 2-sided [-0.56 to 0.32] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Insulin Glargine vs LY2605541 Combined; Test type: Superiority or Other; p = 0.387, Mixed Models Analysis — The statistical significance level is 0.10. P-value is for evening 2-hr postprandial BG; Least Squares Mean Difference (Final) = -0.25, 90% CI 2-sided [-0.73 to 0.23] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Insulin Glargine vs LY2605541 Combined; Test type: Superiority or Other; p = 0.339, Mixed Models Analysis — The statistical significance level is 0.10. P-value is for bed time BG; Least Squares Mean Difference (Final) = -0.29, 90% CI 2-sided [-0.79 to 0.21] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: Insulin Glargine vs LY2605541 Combined; Test type: Superiority or Other; p = 0.676, Mixed Models Analysis — The statistical significance level is 0.10. P-value is for 0300 hours BG; Least Squares Mean Difference (Final) = 0.10, 90% CI 2-sided [-0.30 to 0.50] — [estimate comment as in outcome 1, analysis 1]

7. Secondary Outcome: Daily Basal Insulin Dose at Week 2 and Week 12
Description: LS mean is obtained using MMRM approach, which includes fixed effects of treatment (LY2605541 algorithm 1 and 2, glargine); dose conversion (pre-IA, post-IA); stratification variables (country, baseline daily basal insulin dose group, and baseline HbA1c group); visit; visit and treatment interaction; and a random effect for participant.
Time Frame: Week 2 and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: nanomole per kilogram (nmol/kg)
Arm/Group | Insulin Glargine | LY2605541 Combined
Number analyzed (Participants) | 92 | 188
nanomole per kilogram (nmol/kg)
  Week 2 | 2.45 (0.15) | 3.19 (0.12)
  Week 12: number analyzed (Participants) | 91 | 177
  Week 12 | 2.90 (0.19) | 4.58 (0.15)

8. Secondary Outcome: Percentage of Participants With Hypoglycemia From Baseline Through Week 12
Description: Hypoglycemia episode is defined as any time a participant feels that he/she is experiencing a sign or symptom that is associated with hypoglycemia or has a BG level of ≤3.9 mmol/L (≤70 mg/dL) even if it was not associated with signs, symptoms, or treatment (consistent with current guidelines [ADA 2005]).
Time Frame: Baseline through Week 12
Population: All randomized participants who took at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Insulin Glargine | LY2605541 Combined
Number analyzed (Participants) | 93 | 195
percentage of participants | 63.4 | 54.0
Statistical Analysis 1: Comparison: Insulin Glargine vs LY2605541 Combined; Test type: Superiority or Other; p = 0.162, Fisher Exact — The statistical significance level is 0.10

9. Secondary Outcome: Rate of Hypoglycemia Per 30 Days From Baseline Through Week 12
Description: Hypoglycemia episode is defined as any time a participant feels that he/she is experiencing a sign or symptom that is associated with hypoglycemia or has a BG level of ≤3.9 mmol/L (≤70 mg/dL) even if it was not associated with signs, symptoms, or treatment (consistent with current guidelines [ADA 2005]). Hypoglycemia rate per 30 days is calculated as the number of hypoglycemia/number of days at risk*30.
Time Frame: Baseline through Week 12
Population: All randomized participants who took at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: Number of Hypoglycemia episodes/30 days
Groups:
- LY2605541 Combined: Participants took both LY2605541 and their pre-study insulin for first several days
  Subcutaneous injection of LY2605541 every morning with dose titration based on blood glucose measures for 12 weeks
Arm/Group | Insulin Glargine | LY2605541 Combined
Number analyzed (Participants) | 93 | 195
Number of Hypoglycemia episodes/30 days | 1.52 (2.08) | 1.34 (2.47)
Statistical Analysis 1: Comparison: Insulin Glargine vs LY2605541 Combined; Test type: Superiority or Other; p = 0.804, Negative Binomial Model — The statistical significance level is 0.10

10. Secondary Outcome: Percentage of Participants With Antibody Status Change From Baseline to Week 12 and Week 16
Description: Negative is defined as either 'negative' from lab or percent binding <1.16%. Positive is defined as the percent binding is ≥1.16%. The antibody status change is from negative to positive or positive to negative.
Time Frame: Week 12 and Week 16
Population: All randomized participants who took at least one dose of study drug with both baseline and endpoint antibody measurements.
Measure: Number; unit: percentage of participants
Arm/Group | Insulin Glargine | LY2605541 Algorithm 1 | LY2605541 Algorithm 2
Number analyzed (Participants) | 93 | 98 | 97
percentage of participants
  Week 12 from negative to positive | 2.4 | 4.7 | 2.8
  Week 12 from positive to negative | 2.4 | 0.0 | 1.1
  Week 16 from negative to positive | 2.4 | 4.9 | 3.5
  Week 16 from positive to negative | 2.4 | 0.0 | 1.2

11. Secondary Outcome: Glycemic Variability in Fasting Blood Glucose at Baseline and Week 12
Description: Within-patient glycemic variability was assessed as the standard deviation of fasting blood glucose each day at baseline, and each day between Week 10 and Week 12. LS mean is obtained using MMRM approach, which includes fixed effects of treatment (LY2605541 algorithm 1 and 2, glargine); dose conversion (pre-IA, post-IA); stratification variables (country, baseline daily basal insulin dose group, and baseline HbA1c group); visit; visit and treatment interaction; and a random effect for participant.
Time Frame: Baseline and Week12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: nmol/L
Arm/Group | Insulin Glargine | LY2605541 Combined
Number analyzed (Participants) | 92 | 191
nmol/L
  Baseline | 1.52 (0.11) | 1.51 (0.09)
  Week 12: number analyzed (Participants) | 90 | 177
  Week 12 | 1.23 (0.08) | 1.20 (0.06)
Statistical Analysis 1: Comparison: Insulin Glargine vs LY2605541 Combined; Test type: Superiority or Other; p = 0.937, ANOVA — The statistical significance level is 0.10. P-value is for baseline; Least Squares Mean Difference (Final) = -0.01, 90% CI [-0.16 to 0.14] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Insulin Glargine vs LY2605541 Combined; Test type: Superiority or Other; p = 0.687, Mixed Models Analysis — The statistical significance level is 0.10. P-value is for Week 12; Least Squares Mean Difference (Final) = -0.03, 90% CI 2-sided [-0.16 to 0.10] — [estimate comment as in outcome 1, analysis 1]

12. Secondary Outcome: Pharmacokinetics - Drug (LY2605541) Concentration at Steady State (Css) at Week 12 Endpoint
Description: The drug (LY2605541) concentration at steady state (Css) is calculated from the clearance (Liter/hour) and the final dose of the participants. Clearance was estimated using population-based approaches.
Time Frame: Week 12
Population: Participants who took at least one dose of study drug and had measurements at Week 12.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picomoles per liter (pMol/L)
Arm/Group | LY2605541 Combined
Number analyzed (Participants) | 177
picomoles per liter (pMol/L) | 4258 (70.8)

13. Secondary Outcome: Change From Baseline in Fasting Blood Glucose (FBG) at Week 12 Endpoint - Subgroup Analysis of LY2605541 Dosing Algorithms
Description: FBG is measured by 8-point SMBG profiles, which are measured at morning FBG, midday pre-meal BG, evening pre-meal BG, 2-hour postprandial BG after each of the 3 main meals, bedtime BG, 0300 hours BG. LS mean of the change from baseline to 12 weeks is from MMRM approach. MMRM model includes fixed effects of treatment (LY2605541 algorithm 1, LY2605541 algorithm 2, glargine); stratification variables (country, baseline daily basal insulin dose group, and baseline HbA1c group); visit; visit and treatment interaction; and a random effect for participant.
Time Frame: Baseline, Week 12
Population: All randomized participants who took at least one dose of study drug, excluding those on LY2605541 prior to the changes in the dosing guidance, with non-missing baseline value and at least one non-missing post-baseline value.
Measure: Least Squares Mean (Standard Error); unit: nmol/L
Arm/Group | Insulin Glargine | LY2605541 Algorithm 1 | LY2605541 Algorithm 2
Number analyzed (Participants) | 89 | 70 | 78
nmol/L | -1.82 (0.23) | -2.22 (0.24) | -1.99 (0.23)
Statistical Analysis 1: Comparison: Insulin Glargine vs LY2605541 Algorithm 1; Test type: Superiority or Other; p = 0.159, Mixed Models Analysis — The statistical significance level is 0.10 with no adjustments for multiple comparisons; Least Squares Mean Difference (Final) = -0.40, 90% CI 2-sided [-0.87 to 0.07] — The Least Squares Mean Difference = LY2605541 Algorithm 1 - Insulin Glargine; and 90% confidence interval (CI) = 90% CI of the least squares mean difference
Statistical Analysis 2: Comparison: Insulin Glargine vs LY2605541 Algorithm 2; Test type: Superiority or Other; p = 0.542, Mixed Models Analysis — The statistical significance level is 0.10 with no adjustments for multiple comparisons; Least Squares Mean Difference (Final) = -0.17, 90% CI 2-sided [-0.62 to 0.29] — The Least Squares Mean Difference = LY2605541 Algorithm 2 - Insulin Glargine; and 90% confidence interval (CI) = 90% CI of the least squares mean difference

14. Secondary Outcome: Change From Baseline in HbA1c at Week 12 Endpoint - Subgroup Analysis of LY2605541 Dosing Algorithms
Description: HbA1c is a form of hemoglobin which is measured primarily to identify the average plasma glucose concentration over prolonged periods of time. LS mean of the change from baseline is from MMRM approach. MMRM model includes fixed effects of treatment (LY2605541 algorithm 1, LY2605541 algorithm 2, glargine); stratification variables (country, baseline daily basal insulin dose group); baseline HbA1c; visit; visit and treatment interaction; and a random effect for participant.
Time Frame: Baseline, Week 12
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: percentage of glycated hemoglobin
Arm/Group | Insulin Glargine | LY2605541 Algorithm 1 | LY2605541 Algorithm 2
Number analyzed (Participants) | 91 | 69 | 78
percentage of glycated hemoglobin | -0.65 (0.07) | -0.67 (0.07) | -0.83 (0.07)
Statistical Analysis 1: Comparison: Insulin Glargine vs LY2605541 Algorithm 1; Test type: Superiority or Other; p = 0.880, Mixed Models Analysis — The statistical significance level is 0.10 with no adjustments for multiple comparisons; Least Squares Mean Difference (Final) = -0.01, 90% CI 2-sided [-0.16 to 0.13] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 2: Comparison: Insulin Glargine vs LY2605541 Algorithm 2; Test type: Superiority or Other; p = 0.045, Mixed Models Analysis — The statistical significance level is 0.10 with no adjustments for multiple comparisons; Least Squares Mean Difference (Final) = -0.17, 90% CI 2-sided [-0.32 to -0.03] — [estimate comment as in outcome 13, analysis 2]

15. Secondary Outcome: Percentage of Participants With HbA1c <7.0% and ≤6.5% at Week 12 Endpoint - Subgroup Analysis of LY2605541 Dosing Algorithms
Description: as for outcome 4
Time Frame: Week 12
Population: All randomized participants who took at least one dose of study drug, excluding those on LY2605541 prior to the changes in the dosing guidance, last observation carried forward (LOCF).
Measure: Number; unit: percentage of participants
Arm/Group | Insulin Glargine | LY2605541 Algorithm 1 | LY2605541 Algorithm 2
Number analyzed (Participants) | 91 | 73 | 80
percentage of participants
  HbA1c <7.0% | 48.4 | 57.5 | 50
  HbA1c ≤6.5% | 23.1 | 31.5 | 26.3
Statistical Analysis 1: Comparison: Insulin Glargine vs LY2605541 Algorithm 1; Test type: Superiority or Other; p = 0.273, Fisher Exact — The statistical significance level is 0.10 with no adjustments for multiple comparisons. P-value is for HbA1c <7.0%
Statistical Analysis 2: Comparison: Insulin Glargine vs LY2605541 Algorithm 1; Test type: Superiority or Other; p = 0.287, Fisher Exact — The statistical significance level is 0.10 with no adjustments for multiple comparisons. P-value is for HbA1c ≤6.5%
Statistical Analysis 3: Comparison: Insulin Glargine vs LY2605541 Algorithm 2; Test type: Superiority or Other; p = 0.879, Fisher Exact — The statistical significance level is 0.10 with no adjustments for multiple comparisons. P-value is for HbA1c <7.0%
Statistical Analysis 4: Comparison: Insulin Glargine vs LY2605541 Algorithm 2; Test type: Superiority or Other; p = 0.722, Fisher Exact — The statistical significance level is 0.10 with no adjustments for multiple comparisons. P-value is for HbA1c ≤6.5%

16. Secondary Outcome: Percentage of Participants Who Did Not Experience a Hypoglycemic Episode During Treatment With HbA1c <7.0% and HbA1c ≤6.5% at Week 12 Endpoint - Subgroup Analysis of LY2605541 Dosing Algorithms
Description: HbA1c is a form of hemoglobin which is measured primarily to identify the average plasma glucose concentration over prolonged periods of time. Hypoglycemia episode is defined as any time a participant feels that he/she is experiencing a sign or symptom that is associated with hypoglycemia or has a BG level of ≤3.9 mmol/L (≤70 mg/dL) even if it was not associated with signs, symptoms, or treatment (consistent with current guidelines [ADA 2005]).
Time Frame: Week 12
Population: as for outcome 15
Measure: Number; unit: percentage of participants
Arm/Group | Insulin Glargine | LY2605541 Algorithm 1 | LY2605541 Algorithm 2
Number analyzed (Participants) | 92 | 75 | 83
percentage of participants
  HbA1c <7.0% | 11.96 | 21.33 | 15.66
  HbA1c ≤6.5% | 6.52 | 9.33 | 7.23
Statistical Analysis 1: Comparison: Insulin Glargine vs LY2605541 Algorithm 1; Test type: Superiority or Other; p = 0.139, Fisher Exact — The statistical significance level is 0.10 with no adjustments for multiple comparisons. P-value is for HbA1c <7.0%
Statistical Analysis 2: Comparison: Insulin Glargine vs LY2605541 Algorithm 1; Test type: Superiority or Other; p = 0.569, Fisher Exact — The statistical significance level is 0.10 with no adjustments for multiple comparisons. P-value is for HbA1c ≤6.5%
Statistical Analysis 3: Comparison: Insulin Glargine vs LY2605541 Algorithm 2; Test type: Superiority or Other; p = 0.515, Fisher Exact — The statistical significance level is 0.10 with no adjustments for multiple comparisons. P-value is for HbA1c <7.0%
Statistical Analysis 4: Comparison: Insulin Glargine vs LY2605541 Algorithm 2; Test type: Superiority or Other; p = 1.000, Fisher Exact — The statistical significance level is 0.10 with no adjustments for multiple comparisons. P-value is for HbA1c ≤6.5%

17. Secondary Outcome: 8-Point Self-Monitored Blood Glucose (SMBG) Measures at Week 12 Endpoint - Subgroup Analysis of LY2605541 Dosing Algorithms
Description: 8-point SMBG profiles are measured at morning FBG, midday pre-meal BG, evening pre-meal BG, 2-hour postprandial BG after each of the 3 main meals, bedtime BG, 0300 hours BG. LS mean is obtained using MMRM approach, which includes fixed effects of treatment (LY2605541 algorithm 1, LY2605541 algorithm 2, glargine); stratification variables (country, baseline daily basal insulin dose group, and baseline HbA1c group); visit; visit and treatment interaction; and a random effect for participant.
Time Frame: Week 12
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: nmol/L
Arm/Group | Insulin Glargine | LY2605541 Algorithm 1 | LY2605541 Algorithm 2
Number analyzed (Participants) | 92 | 78 | 83
nmol/L
  Morning pre-meal BG: number analyzed (Participants) | 89 | 70 | 78
  Morning pre-meal BG | 6.76 (0.19) | 7.02 (0.21) | 6.62 (0.20)
  Morning 2-hr postprandial BG: number analyzed (Participants) | 87 | 70 | 76
  Morning 2-hr postprandial BG | 9.31 (0.27) | 9.05 (0.29) | 8.48 (0.28)
  Midday Pre-meal BG: number analyzed (Participants) | 89 | 70 | 77
  Midday Pre-meal BG | 7.29 (0.26) | 7.22 (0.27) | 6.60 (0.26)
  Midday 2-hr postprandial BG: number analyzed (Participants) | 88 | 70 | 76
  Midday 2-hr postprandial BG | 9.36 (0.25) | 8.96 (0.27) | 9.09 (0.26)
  Evening Pre-meal BG: number analyzed (Participants) | 89 | 69 | 78
  Evening Pre-meal BG | 7.79 (0.25) | 7.64 (0.27) | 7.64 (0.25)
  Evening 2-hr postprandial BG: number analyzed (Participants) | 89 | 70 | 77
  Evening 2-hr postprandial BG | 9.64 (0.26) | 9.14 (0.28) | 9.22 (0.27)
  Bed time BG: number analyzed (Participants) | 80 | 62 | 69
  Bed time BG | 9.13 (0.27) | 8.86 (0.29) | 8.43 (0.28)
  0300 hours BG: number analyzed (Participants) | 89 | 68 | 73
  0300 hours BG | 7.10 (0.22) | 7.34 (0.24) | 6.82 (0.23)
Statistical Analysis 1: Comparison: Insulin Glargine vs LY2605541 Algorithm 1; Test type: Superiority or Other; p = 0.305, Mixed Models Analysis — The statistical significance level is 0.10 with no adjustments for multiple comparisons. P-value is for morning pre-meal BG; Least Squares Mean Difference (Final) = 0.26, 90% CI 2-sided [-0.16 to 0.67] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 2: Comparison: Insulin Glargine vs LY2605541 Algorithm 2; Test type: Superiority or Other; p = 0.571, Mixed Models Analysis — [p-value comment as in outcome 17, analysis 1]; Least Squares Mean Difference (Final) = -0.14, 90% CI 2-sided [-0.54 to 0.26] — [estimate comment as in outcome 13, analysis 2]
Statistical Analysis 3: Comparison: Insulin Glargine vs LY2605541 Algorithm 1; Test type: Superiority or Other; p = 0.454, Mixed Models Analysis — The statistical significance level is 0.10 with no adjustments for multiple comparisons. P-value is for morning 2-hr postprandial BG; Least Squares Mean Difference (Final) = -0.26, 90% CI [-0.85 to 0.32] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 4: Comparison: Insulin Glargine vs LY2605541 Algorithm 2; Test type: Superiority or Other; p = 0.016, Mixed Models Analysis — [p-value comment as in outcome 17, analysis 3]; Least Squares Mean Difference (Final) = -0.83, 90% CI 2-sided [-1.40 to -0.26] — [estimate comment as in outcome 13, analysis 2]
Statistical Analysis 5: Comparison: Insulin Glargine vs LY2605541 Algorithm 1; Test type: Superiority or Other; p = 0.838, Mixed Models Analysis — The statistical significance level is 0.10 with no adjustments for multiple comparisons. P-value is for midday pre-meal BG; Least Squares Mean Difference (Final) = -0.07, 90% CI [-0.61 to 0.48] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 6: Comparison: Insulin Glargine vs LY2605541 Algorithm 2; Test type: Superiority or Other; p = 0.033, Mixed Models Analysis — [p-value comment as in outcome 17, analysis 5]; Least Squares Mean Difference (Final) = -0.69, 90% CI 2-sided [-1.22 to -0.16] — [estimate comment as in outcome 13, analysis 2]
Statistical Analysis 7: Comparison: Insulin Glargine vs LY2605541 Algorithm 1; Test type: Superiority or Other; p = 0.229, Mixed Models Analysis — The statistical significance level is 0.10 with no adjustments for multiple comparisons. P-value is for midday 2-hr postprandial BG; Least Squares Mean Difference (Final) = -0.40, 90% CI 2-sided [-0.95 to 0.15] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 8: Comparison: Insulin Glargine vs LY2605541 Algorithm 2; Test type: Superiority or Other; p = 0.412, Mixed Models Analysis — [p-value comment as in outcome 17, analysis 7]; Least Squares Mean Difference (Final) = -0.27, 90% CI 2-sided [-0.80 to 0.27] — [estimate comment as in outcome 13, analysis 2]
Statistical Analysis 9: Comparison: Insulin Glargine vs LY2605541 Algorithm 1; Test type: Superiority or Other; p = 0.642, Mixed Models Analysis — The statistical significance level is 0.10 with no adjustments for multiple comparisons. P-value is for evening pre-meal BG; Least Squares Mean Difference (Final) = -0.15, 90% CI 2-sided [-0.68 to 0.38] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 10: Comparison: Insulin Glargine vs LY2605541 Algorithm 2; Test type: Superiority or Other; p = 0.614, Mixed Models Analysis — [p-value comment as in outcome 17, analysis 9]; Least Squares Mean Difference (Final) = -0.16, 90% CI 2-sided [-0.67 to 0.36] — [estimate comment as in outcome 13, analysis 2]
Statistical Analysis 11: Comparison: Insulin Glargine vs LY2605541 Algorithm 1; Test type: Superiority or Other; p = 0.147, Mixed Models Analysis — The statistical significance level is 0.10 with no adjustments for multiple comparisons. P-value is for evening 2-hr postprandial BG; Least Squares Mean Difference (Final) = -0.50, 90% CI 2-sided [-1.07 to 0.07] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 12: Comparison: Insulin Glargine vs LY2605541 Algorithm 2; Test type: Superiority or Other; p = 0.210, Mixed Models Analysis — [p-value comment as in outcome 17, analysis 11]; Least Squares Mean Difference (Final) = -0.42, 90% CI 2-sided [-0.98 to 0.13] — [estimate comment as in outcome 13, analysis 2]
Statistical Analysis 13: Comparison: Insulin Glargine vs LY2605541 Algorithm 1; Test type: Superiority or Other; p = 0.438, Mixed Models Analysis — The statistical significance level is 0.10 with no adjustments for multiple comparisons. P-value is for bed time BG; Least Squares Mean Difference (Final) = -0.28, 90% CI 2-sided [-0.86 to 0.31] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 14: Comparison: Insulin Glargine vs LY2605541 Algorithm 2; Test type: Superiority or Other; p = 0.043, Mixed Models Analysis — The statistical significance level is 0.10 with no adjustments for multiple comparisons. P-value is for bed time BG; Least Squares Mean Difference (Final) = -0.70, 90% CI 2-sided [-1.28 to -0.13] — [estimate comment as in outcome 13, analysis 2]
Statistical Analysis 15: Comparison: Insulin Glargine vs LY2605541 Algorithm 1; Test type: Superiority or Other; p = 0.403, Mixed Models Analysis — The statistical significance level is 0.10 with no adjustments for multiple comparisons. P-value is for 0300 hours BG; Least Squares Mean Difference (Final) = 0.24, 90% CI 2-sided [-0.23 to 0.72] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 16: Comparison: Insulin Glargine vs LY2605541 Algorithm 2; Test type: Superiority or Other; p = 0.314, Mixed Models Analysis — The statistical significance level is 0.10 with no adjustments for multiple comparisons. P-value is for 0300 hours BG; Least Squares Mean Difference (Final) = -0.29, 90% CI 2-sided [-0.75 to 0.18] — [estimate comment as in outcome 13, analysis 2]

18. Secondary Outcome: Daily Basal Insulin Dose at Week 2 and Week 12 - Subgroup Analysis of LY2605541 Dosing Algorithms
Description: LS mean is obtained using MMRM approach, which includes fixed effects of treatment (LY2605541 algorithm 1, LY2605541 algorithm 2, glargine); stratification variables (country, baseline daily basal insulin dose group, and baseline HbA1c group); visit; visit and treatment interaction; and a random effect for participant.
Time Frame: Week 2 and Week 12
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: nmol/kg
Arm/Group | Insulin Glargine | LY2605541 Algorithm 1 | LY2605541 Algorithm 2
Number analyzed (Participants) | 92 | 76 | 81
nmol/kg
  Week 2 | 2.62 (0.13) | 3.23 (0.13) | 3.64 (0.13)
  Week 12: number analyzed (Participants) | 91 | 70 | 78
  Week 12 | 3.15 (0.16) | 4.58 (0.17) | 5.26 (0.17)

19. Secondary Outcome: Percentage of Participants With Hypoglycemia From Baseline Through Week 12 - Subgroup Analysis of LY2605541 Dosing Algorithms
Description: as for outcome 8
Time Frame: Baseline through Week 12
Population: All randomized participants who took at least one dose of study drug, excluding those on LY2605541 prior to the changes in the dosing guidance.
Measure: Number; unit: percentage of participants
Arm/Group | Insulin Glargine | LY2605541 Algorithm 1 | LY2605541 Algorithm 2
Number analyzed (Participants) | 93 | 80 | 83
percentage of participants | 63.4 | 47.5 | 54.2
Statistical Analysis 1: Comparison: Insulin Glargine vs LY2605541 Algorithm 1; Test type: Superiority or Other; p = 0.046, Fisher Exact — The statistical significance level is 0.10 with no adjustments for multiple comparisons
Statistical Analysis 2: Comparison: LY2605541 Algorithm 2; Test type: Superiority or Other; p = 0.224, Fisher Exact — The statistical significance level is 0.10 with no adjustments for multiple comparisons

20. Secondary Outcome: Rate of Hypoglycemia Per 30 Days From Baseline Through Week 12 - Subgroup Analysis of LY2605541 Dosing Algorithms
Description: as for outcome 9
Time Frame: Baseline through Week 12
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: Number of Hypoglycemia episodes/30 days
Arm/Group | Insulin Glargine | LY2605541 Algorithm 1 | LY2605541 Algorithm 2
Number analyzed (Participants) | 93 | 80 | 83
Number of Hypoglycemia episodes/30 days | 1.52 (2.08) | 1.25 (2.27) | 1.27 (2.20)
Statistical Analysis 1: Comparison: Insulin Glargine vs LY2605541 Algorithm 1; Test type: Superiority or Other; p = 0.561, Negative Binomial Model — The statistical significance level is 0.10 with no adjustments for multiple comparisons
Statistical Analysis 2: Comparison: Insulin Glargine vs LY2605541 Algorithm 2; Test type: Superiority or Other; p = 0.518, Negative Binomial Model — The statistical significance level is 0.10 with no adjustments for multiple comparisons

21. Secondary Outcome: Glycemic Variability in Fasting Blood Glucose at Baseline and Week 12 - Subgroup Analysis of LY2605541 Dosing Algorithms
Description: Within-patient glycemic variability was assessed as the standard deviation of fasting blood glucose each day at baseline, and each day between Week 10 and Week 12. LS mean is obtained using MMRM approach, which includes fixed effects of treatment (LY2605541 algorithm 1, LY2605541 algorithm 2, glargine); stratification variables (country, baseline daily basal insulin dose group, and baseline HbA1c group); visit; interaction between visit and treatment; and a random effect for participant.
Time Frame: Baseline and Week 12
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: nmol/L
Arm/Group | Insulin Glargine | LY2605541 Algorithm 1 | LY2605541 Algorithm 2
Number analyzed (Participants) | 92 | 77 | 83
nmol/L
  Baseline | 1.43 (0.07) | 1.40 (0.08) | 1.42 (0.07)
  Week 12: number analyzed (Participants) | 90 | 70 | 78
  Week 12 | 1.17 (0.07) | 1.16 (0.08) | 1.07 (0.07)
Statistical Analysis 1: Comparison: Insulin Glargine vs LY2605541 Algorithm 1; Test type: Superiority or Other; p = 0.938, ANOVA — The statistical significance level is 0.10 with no adjustments for multiple comparisons. P-value is for baseline; Least Squares Mean Difference (Final) = -0.01, 90% CI 2-sided [-0.20 to 0.18] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 2: Comparison: Insulin Glargine vs LY2605541 Algorithm 2; Test type: Superiority or Other; p = 0.972, ANOVA — The statistical significance level is 0.10 with no adjustments for multiple comparisons. P-value is for baseline; Least Squares Mean Difference (Final) = 0.00, 90% CI 2-sided [-0.18 to 0.19] — [estimate comment as in outcome 13, analysis 2]
Statistical Analysis 3: Comparison: Insulin Glargine vs LY2605541 Algorithm 1; Test type: Superiority or Other; p = 0.927, Mixed Models Analysis — The statistical significance level is 0.10 with no adjustments for multiple comparisons. P-value is for Week 12; Least Squares Mean Difference (Final) = -0.01, 90% CI 2-sided [-0.16 to 0.15] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 4: Comparison: Insulin Glargine vs LY2605541 Algorithm 2; Test type: Superiority or Other; p = 0.293, Mixed Models Analysis — The statistical significance level is 0.10 with no adjustments for multiple comparisons. P-value is for Week 12; Least Squares Mean Difference (Final) = -0.10, 90% CI 2-sided [-0.25 to 0.05] — [estimate comment as in outcome 13, analysis 2]

ADVERSE EVENTS:
Groups:
- LY2605541 Dosing Algorithm 1; LY2605541 Dosing Algorithm 2: subcutaneous injection of LY2605541 every morning with dose titration based on blood glucose measures for 12 weeks
Arm/Group | LY2605541 Dosing Algorithm 1 | LY2605541 Dosing Algorithm 2 | Insulin Glargine
Serious Adverse Events (participants affected / at risk) | 4/98 | 1/98 | 2/93
Other Adverse Events (participants affected / at risk) | 44/98 | 47/98 | 45/93
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY2605541 Dosing Algorithm 1 (N=98) | LY2605541 Dosing Algorithm 2 (N=98) | Insulin Glargine (N=93)
Angina unstable (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Foreign body (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY2605541 Dosing Algorithm 1 (N=98) | LY2605541 Dosing Algorithm 2 (N=98) | Insulin Glargine (N=93)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 3 (3) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 3 (3) | 3 (3)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2)
Asthenia (General disorders) | 2 (2) | 0 (0) | 0 (0)
Fatigue (General disorders) | 2 (2) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1) | 2 (2)
Influenza (Infections and infestations) | 3 (3) | 2 (2) | 0 (0)
Nasopharyngitis (Infections and infestations) | 3 (3) | 6 (6) | 5 (6)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 3 (3) | 3 (3)
Urinary tract infection (Infections and infestations) | 0 (0) | 3 (3) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 2 (2) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 2 (3) | 0 (0) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 0 (0) | 2 (2)
Abnormal loss of weight (Metabolism and nutrition disorders) | 2 (2) | 4 (4) | 1 (1)
Abnormal weight gain (Metabolism and nutrition disorders) | 0 (0) | 2 (3) | 3 (3)
Dyslipidaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Underweight (Metabolism and nutrition disorders) | 1 (1) | 4 (4) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (3) | 4 (4)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 3 (3) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 4 (4) | 2 (2) | 4 (6)
Insomnia (Psychiatric disorders) | 2 (6) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days